CLINICAL TRIAL: NCT00716066
Title: High-Dose Immunosuppressive Therapy Using Carmustine, Etoposide, Cytarabine, and Melphalan (BEAM) + Thymoglobulin Followed by Syngeneic or Autologous Hematopoietic Cell Transplantation for Patients With Autoimmune Neurologic Diseases
Brief Title: Autologous Stem Cell Transplant for Neurologic Autoimmune Diseases
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2260.00; NCI-2010-00403 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2260.00 (Other: Fred Hutch/University of Washington Cancer Consortium); RG9213030 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2008-07-15; First posted 2008-07-16 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Autoimmune Disease; Neurologic Autoimmune Disease; Autologous Transplant Autoimmune; Multiple Sclerosis Transplant; MS Stem Cell Transplant; Multiple Sclerosis Stem Cell Transplant; Stiff Person Syndrome; HCT for Neurologic Autoimmune Disorders; CIDP Transplant; Myasthenia Gravis Transplant; Autoimmune Nervous System Disorder; Central Nervous System Vasculitis; Cerebellar Degeneration; Chronic Inflammatory Demyelinating Polyneuropathy; Lambert Eaton Myasthenic Syndrome; Myasthenia Gravis; Neuromyelitis Optica; Opsoclonus Myoclonus Syndrome; Rasmussen Subacute Encephalitis
Keywords: neurologic autoimmune disease; autologous transplant autoimmune; multiple sclerosis transplant; MS stem cell transplant; multiple sclerosis stem cell transplant; Stiff Person Syndrome; HCT for neurologic autoimmune disorders; CIDP transplant; myasthenia gravis transplant
MeSH Terms: conditions — Autoimmune Diseases; Autoimmune Diseases of the Nervous System; Stiff-Person Syndrome; Vasculitis, Central Nervous System; Polyradiculoneuropathy, Chronic Inflammatory Demyelinating; Lambert-Eaton Myasthenic Syndrome; Myasthenia Gravis; Neuromyelitis Optica; Opsoclonus-Myoclonus Syndrome; Rasmussen subacute encephalitis | interventions — Antilymphocyte Serum; thymoglobulin; Carmustine; carmustine, poliferprosan 20 drug combination; Cytarabine; Etoposide; Melphalan; Peripheral Blood Stem Cell Transplantation; Prednisone; deltacortene; prednylidene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (immunosuppressive therapy followed by transplant) (Experimental): Patients receive carmustine IV on day -6, etoposide IV and cytarabine IV BID on days -5 to -2, melphalan IV on day -1 and antithymocyte globulin IV on days -2 and -1. Patients then undergo autologous or syngeneic stem cell transplant on day 0. Patients also receive prednisone PO QD on days 7-21, followed by 2 week taper.
  Interventions: Biological: Anti-Thymocyte Globulin; Procedure: Autologous Hematopoietic Stem Cell Transplantation; Drug: Carmustine; Drug: Cytarabine; Drug: Etoposide; Other: Laboratory Biomarker Analysis; Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Prednisone; Procedure: Syngeneic Bone Marrow Transplantation

INTERVENTIONS:
Biological: Anti-Thymocyte Globulin — Given IV
  Other Names: Antithymocyte Globulin; Antithymocyte Serum; ATG; ATGAM; ATS; Thymoglobulin
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous or syngeneic stem cell transplantation
  Other Names: Autologous Stem Cell Transplantation
Drug: Carmustine — Given IV
  Other Names: BCNU; Becenum; Becenun; BiCNU; Bis(chloroethyl) Nitrosourea; Bis-Chloronitrosourea; Carmubris; Carmustin; Carmustinum; FDA 0345; Gliadel; N,N'-Bis(2-chloroethyl)-N-nitrosourea; Nitrourean; Nitrumon; SK 27702; SRI 1720; WR-139021; 154-93-8
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosar-U; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453; 147-94-4
Drug: Etoposide — Given IV
  Other Names: Demethyl Epipodophyllotoxin Ethylidine Glucoside; EPEG; Lastet; Toposar; Vepesid; VP 16-213; VP-16; VP-16-213; 33419-42-0
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine Mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813; 148-82-3
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous or syngeneic stem cell transplantation
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone; 53-03-2
Procedure: Syngeneic Bone Marrow Transplantation — Undergo syngeneic bone marrow transplantation

SUMMARY:
This phase II trial studies the side effects and how well carmustine, etoposide, cytarabine and melphalan together with antithymocyte globulin before a stem cell transplant works in treating patients with autoimmune neurologic disease that did not respond to previous therapy. In autoimmune neurological diseases, the patient's own immune system 'attacks' the nervous system which might include the brain/spinal cord and/or the peripheral nerves. Giving high-dose chemotherapy, including carmustine, etoposide, cytarabine, melphalan, and antithymocyte globulin, before a stem cell transplant weakens the immune system and may help stop the immune system from 'attacking' a patient's nervous system. When the patient's own (autologous) stem cells are infused into the patient they help the bone marrow make red blood cells, white blood cells, and platelets so the blood counts can improve.

DETAILED DESCRIPTION:
OUTLINE:

Patients receive carmustine intravenously (IV) on day -6, etoposide IV and cytarabine IV twice daily (BID) on days -5 to -2, melphalan IV on day -1, and antithymocyte globulin IV on days -2 and -1. Patients then undergo autologous or syngeneic stem cell transplant on day 0. Patients also receive prednisone orally (PO) once daily (QD) on days 7-21, followed by 2 week taper.

After completion of study treatment, patients are followed up at 3 months, 1 year, and then annually thereafter for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an autoimmune disorder of the central or peripheral nervous system will be eligible; this will include:

  * Primary Central Nervous System (CNS) vasculitis
  * Rasmussen's encephalitis
  * Autoimmune peripheral neuropathy (anti-Hu [Anna-1], anti-GM1 [GD1b], anti-MAG, anti-ganglioside, anti-sulfatide)
  * Autoimmune cerebellar degeneration
  * Gait Ataxia with Late age Onset Polyneuropathy (GALOP)
  * Stiff Person Syndrome
  * Chronic Inflammatory Demyelinating Polyneuropathy
  * Myasthenia Gravis
  * Lambert-Eaton myasthenic syndrome
  * Human T-cell lymphotropic virus (HTLV)-1-associated myelopathy (HAM) / tropical spastic paraparesis (TSP)
  * Opsoclonus/myoclonus (anti-Ri)
  * Neuromyelitis optica
  * Multiple sclerosis
  * Other central or peripheral nervous system autoimmune diseases as approved by study neurologists and the Fred Hutchinson Cancer Research Center (FHCRC) faculty at Patient Care Conference (PCC)
* Patients must satisfy the criteria for a diagnosis of one of the severe neurological autoimmune disorders outlined
* Patients age =< 70 years
* Evidence of disease activity as outlined (e.g. gadolinium enhancement on magnetic resonance imaging of the brain or clinical progression)
* Patients must have failed at least 2 lines of standard therapy as outlined for the specific diseases
* DONOR: Sibling of any patient enrolled on this protocol proven by ABO typing, human leukocyte antigen (HLA) typing and variable number tandem repeat (VNTR) analysis to be syngeneic with the patient (e.g. identical twin)
* DONOR: Willing to undergo multiple apheresis procedures (except donors < 12 years who will undergo bone marrow harvests)

Exclusion Criteria:

* Age >= 71 years
* Pregnancy or expressed plans to become pregnant within 1 year of the procedure
* Patients who are serologically positive for human immunodeficiency virus (HIV)
* Patients with pulmonary, cardiac, hepatic or renal impairment that would limit their ability to receive cytoreductive therapy and compromise their survival; this should include patients with any of the following:

  * Severe pulmonary dysfunction associated with a carbon monoxide diffusing capacity (DLCO) (corrected for hemoglobin) < 60%, or requires supplemental oxygen; patients who are unable to perform pulmonary function test (because of underlying disease) will be excluded if the oxygen saturation is < 92% on room air
  * Uncontrolled malignant arrhythmias, or clinical evidence of congestive heart failure (New York class III-IV) or ejection fraction < 50%
  * Renal disease with estimated glomerular filtration rate (GFR) by creatinine clearance or iothalamate clearance < 50 ml/min/1.73 m^2 body surface area
  * Serum glutamate pyruvate transaminase (SGPT)/aspartate aminotransferase (AST) > 3 times normal or direct bilirubin greater than 2.5 mg/dL on two repeated tests
* Active uncontrolled infection
* Demonstrated lack of compliance with prior medical care
* Patients whose life expectancy is limited by illness other than their neurological condition
* Patients with evidence of myelodysplasia
* Active malignancy (excluding localized squamous cell or basal cell carcinoma of the skin)
* DONOR: Inadequate documentation that donor and recipient are syngeneic
* DONOR: Donors who do not fulfill criteria as apheresis donors as established by institutional guidelines
* DONOR: Concordant for autoimmune neurological disease(s) as determined by neurological evaluation

Max Age: 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2008-06; Primary Completion 2025-12-30 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of grades 4-5 regimen-related toxicity | Up to 1 year post-transplant
  Assessed by the Regimen Related Toxicity Scale. Using the National Cancer Institute Common Terminology Criteria for Adverse Events version 3.0. The development of a grade 4 to 5 toxicity of any of the included major organ systems within the first 365 days after transplant will be defined as regimen-related toxicity.

SECONDARY OUTCOMES:
Transplant-related mortality | Within 100 days post-transplant
  Defined as death within the first 100 days of transplant due to transplant-related complications.
Disease responses | Up to 5 years
  Assessed by clinical, laboratory and radiologic evaluation
Engraftment kinetics | Over first 60 days post-transplant
  Monitored for engraftment kinetics of granulocytes, platelets and red cells post-transplant.
Number of subjects achieving greater than or equal to 4.0 x 10^6 CD34+ cells/kg, after up to two peripheral blood stem cell mobilizations | Baseline to post mobilization, assessed up to 20 days after starting final mobilization (up to two mobilizations)
  Efficacy of peripheral blood stem cell mobilization as evaluated by total number of harvested CD34+cells/kg, for autologous transplant.
Number of subjects with an exacerbation of autoimmune disease symptoms secondary to G-CSF (filgrastim) during peripheral blood stem cell mobilization | Baseline to post mobilization, assessed up to 20 days after starting final mobilization (up to two mobilizations)
  Subjects are evaluated by standardized clinical neurologic tests specific to autoimmune disease type.

CONTACTS AND LOCATIONS:
Overall Officials: Leona Holmberg, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington